CLINICAL TRIAL: NCT04992728
Title: Quantitative Diffusion MRI for Prostate Cancer Detection and Monitoring
Brief Title: Prostate Assessment with Restriction Spectrum Imaging (RSI) MRI
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tyler Seibert, Assistant Professor of Medicine, University of California, San Diego
Other Study IDs: 805338
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Male Prostate Patients: Adult male patients with fair to good performance status and who (1) have undergone an MRI of the prostate for suspected or known prostate cancer and/or (2) are planning to undergo radical prostatectomy for prostate cancer.
  Interventions: Other: Restricted Spectrum Magnetic Resonance Imagining

INTERVENTIONS:
Other: Restricted Spectrum Magnetic Resonance Imagining — Restriction Spectrum Magnetic Resonance Imaging (RS-MRI), which uses magnetism instead of x-rays to build up a picture of the inside of the body. The scan is completely painless but can be rather noisy and requires the patient to lie very still inside the center of a large, doughnut-shaped magnet for approximately 30-60 minutes complete the imaging.
  Other Names: RSI MRI; Diffusion MRI

SUMMARY:
This single-center study will enroll 40 male participants to complete 2 diffusion magnetic resonance images within 30 days of each other.

DETAILED DESCRIPTION:
Participants will undergo prostate MRI using a range of b-values and echo times. 40 participants will be invited to complete two such scans within 30 days of each other to evaluate reliability across time. Several advanced MRI models will be applied to the data, and the models will be assessed for accurate prediction of grade group ≥2 prostate cancer on histopathology, obtained through routine clinical care. We hypothesize that advanced, multi-compartment dMRI will yield a reliable, quantitative metric that is superior to standard ADC for detection of csPCa.

RSI is a multicompartment model of diffusion MRI that uses data acquired at multiple b-values to distinguish varied diffusion speeds (restricted intracellular, hindered extracellular, and approximately free diffusion). The relative contributions of each compartment are estimated for each voxel in the imaging field of view. RSI cellularity index is a normalized parameter reflecting the contribution of very slow diffusion that is associated with tumor cellularity.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged ≥18 years, with histologically confirmed adenocarcinoma of the prostate
* Has already undergone prostate MRI and/or scheduled to undergo clinically indicated radical prostatectomy (to permit whole-mount histopathology correlation).
* Intended treatment and follow-up according to standard of care for prostate cancer
* In good general health as evidenced by medical history and ECOG performance status 0-2
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Prior treatment for prostate cancer (cryotherapy, high frequency focused ultrasound, prostatectomy)
* Hip prosthesis
* Contraindication to MRI, per institutional requirements
* Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biological males with intact prostate
Study Population: Adult male patients with fair to good performance status and who (1) have undergone an MRI of the prostate for suspected or known prostate cancer and/or (2) are planning to undergo radical prostatectomy for prostate cancer.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Detection of grade group ≥2 prostate cancer on histopathology | 30 days
  To determine an optimal quantitative dMRI technique for csPCa detection, we will implement an expanded dMRI protocol that will permit exploration of six different approaches, each with published evidence of advantages over conventional ADC. Accuracy will be evaluated using histopathology as the gold standard.

SECONDARY OUTCOMES:
Inter-scan reliability | 30 days
  Reliability is a critical feature of quantitative imaging biomarkers. Prostate MRI is known to vary with physiologic conditions, such as bowel activity, bowel/bladder filling, and recency of ejaculation(5). Patients planning to undergo prostatectomy (to permit whole-mount histopathology correlation) will be invited to consent to a second MRI scan on a different date, within approximately 30 days of the first scan (to avoid meaningful change in any tumor). The across-date reproducibility coefficient will be calculated for each metric

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Seibert, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No